CLINICAL TRIAL: NCT01317771
Title: Analysis of the Fixation of the Proximal Long Head of the Biceps Tendon
Brief Title: Analysis of the Fixation of the Proximal Biceps Tendon
Status: Withdrawn | Type: Observational
Why Stopped: PI decided to not activate
Sponsor: West Penn Allegheny Health System (Other)
Responsible Party: Principal Investigator, Carmen Latona, PI, West Penn Allegheny Health System
Other Study IDs: RC-5202
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Disorder of Tendon of Biceps
Keywords: Proximal Biceps Pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Proximal Biceps Tendon Tenodesis
  Interventions: Procedure: Open proximal biceps tendon tenodesis with an EndoButton

INTERVENTIONS:
Procedure: Open proximal biceps tendon tenodesis with an EndoButton — Surgical fixation for bicipital pathology

SUMMARY:
Ten randomly selected patients that have undergone an open proximal biceps tendon tenodesis with an EndoButton for bicipital pathology with Christopher Schmidt, MD, will be asked to participate in the study. The study will assess the tendon healing to bone through magnetic resonance imaging (MRI). Individuals will also be asked to fill a visual analog scale (VAS) pain and disability of the arm shoulder and hand (DASH) assessment tools. The variables for our objective will include age, hand dominance, gender and chronicity of symptoms prior to surgery, and other related surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Undergone open subpectoral proximal biceps tenodesis with the EndoButton

Exclusion Criteria:

* No history of surgery or disability in the contra-lateral extremity
* Not a member of a legally restricted group or protected population
* No prior surgery or further surgery on the extremity of interest
* No condition preventing the individual from undergoing a MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research study will collect the MRI and questionnaire data from 10 subjects that have undergone a subpectoral proximal biceps tendon tenodesis using the EndoButton.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-03-11 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Schmidt, MD, Principal Investigator — WPAHS
Locations (1):
- Allegheny Imaging of McCandless, Pittsburgh, Pennsylvania, United States